CLINICAL TRIAL: NCT00000157
Title: Randomized Trial of Aspirin and Cataracts in U.S. Physicians
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: NEI-59
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
To determine whether 325 mg of aspirin taken on -alternate days reduces the risk of developing cataract among male U.S. physicians who were aged 40 to 84 in 1982.

To identify potential risk factors for cataract development, such as age, blood pressure, blood cholesterol, height, diabetes, medication use, and history of previous eye trauma or surgery.

DETAILED DESCRIPTION:
Cataract is one of the most common causes of impaired vision as well as the third leading cause of blindness in the United States. Cataract surgery is one of the safest and most successful of all operations. The National Eye Institute has estimated that if the progression of cataract could be slowed enough to delay the need for surgery by even 10 years, the current annual number could be reduced by 45 percent.

Little is known about the relative importance of various potential risk factors in the development of cataract. Most current information on risk factors has come from anecdotal reports or from relatively small case-control studies. One major project, the Framingham Eye Study, has identified several factors that were significantly associated with subsequent cataract formation, including diabetes and dietary factors. Diabetes has long been thought to increase the risk of developing cataract.

Recently, aspirin has been proposed as a drug that can prevent cataract formation or slow its progression. Aspirin may affect tryptophan levels in patients with cataract, or it may inhibit aldose reductase, an enzyme associated with the development of diabetic cataract. Thus, data from this study sought to determine whether one 325-mg aspirin tablet, taken on alternate days, protects against cataract formation. The data also sought to reveal other additional cataract risk factors that emerge after simultaneous controlling for other variables.

The other primary objective of this trial was to assess the antioxidant effects of beta-carotene (50 mg on alternate days) on cataract development. In addition, factors that have been suggested to be cataractogenic were assessed in prospective cohort studies. These factors included age, blood pressure, blood cholesterol, height, diabetes, medication use, cigarette smoking, and history of previous eye trauma or surgery. In addition, the possible associations between history of vitamin E and selenium intake and cataract were explored.

This trial was part of the Physicians Health Study, an ongoing, randomized, placebo-controlled clinical trial of aspirin in the prevention of cardiovascular mortality and of beta-carotene in the prevention of cancer. Following randomization, each of the 22,071 physicians enrolled was assigned to one of four groups to take either aspirin or its placebo and beta-carotene or its placebo. Follow-up questionnaires were sent 6 and 12 months after randomization and every 12 months thereafter. The randomized aspirin component of the trial was terminated early (January 1988), after an average followup of approximately 5 years, because of a statistically extreme 44 percent reduced risk of a first myocardial infarction in the aspirin group.

Since this study is conducted by mail among physicians nationwide, examinations cannot be performed on all patients to determine when they have reached an end point. Reported diagnoses of cataract are confirmed by medical record review. The primary analysis will be of incidence of cataract in the aspirin and placebo groups. In addition, the Cox proportional hazards model will be used to determine whether there is a difference in time to cataract diagnosis between the two groups. It has been postulated that the potent antioxidant properties of beta-carotene might make it effective in preventing cataract development. The investigators will thus determine whether there is a difference in the numbers of cataracts between the beta-carotene/placebo groups and the aspirin/placebo groups.

ELIGIBILITY:
The study population consisted of 22,071 male U.S. physicians, aged 40 to 84 years in 1982, with no history of myocardial infarction, cancer, kidney disease, renal disease, or any other contraindication to the use of aspirin or beta-carotene, including regular use of corticosteroids.

Ages: 40 Years to 84 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1982-04; Study Completion 1988-01 (Actual)

REFERENCES:
- [Background] Seddon JM, Christen WG, Manson JE, Buring JE, Sperduto RD, Hennekens CH. Low-dose aspirin and risks of cataract in a randomized trial of US physicians. Arch Ophthalmol. 1991 Feb;109(2):252-5. doi: 10.1001/archopht.1991.01080020098052. PMID 1993037
- [Background] Christen WG, Manson JE, Seddon JM, Glynn RJ, Buring JE, Rosner B, Hennekens CH. A prospective study of cigarette smoking and risk of cataract in men. JAMA. 1992 Aug 26;268(8):989-93. PMID 1501324
- [Background] Christen WG, Glynn RJ, Seddon JM, Manson JE, Buring JE, Hennekens CH. Confirmation of self-reported cataract in the Physicians' Health Study. Ophthalmic Epidemiol. 1994 Jun;1(2):85-91. doi: 10.3109/09286589409052364. PMID 8790615
- [Background] Manson JE, Christen WG, Seddon JM, Glynn RJ, Hennekens CH. A prospective study of alcohol consumption and risk of cataract. Am J Prev Med. 1994 May-Jun;10(3):156-61. PMID 7917442
- [Background] Seddon JM, Christen WG, Manson JE, LaMotte FS, Glynn RJ, Buring JE, Hennekens CH. The use of vitamin supplements and the risk of cataract among US male physicians. Am J Public Health. 1994 May;84(5):788-92. doi: 10.2105/ajph.84.5.788. PMID 8179050
- [Background] Glynn RJ, Christen WG, Manson JE, Bernheimer J, Hennekens CH. Body mass index. An independent predictor of cataract. Arch Ophthalmol. 1995 Sep;113(9):1131-7. doi: 10.1001/archopht.1995.01100090057023. PMID 7661746